CLINICAL TRIAL: NCT06404333
Title: A Randomized Trial to Assess the Safety, Pharmacokinetics, Acceptability, and Efficacy of Pediatric Oral Ivermectin in Scabies Infected Children Weighing 5 to Less Than 15 Kilograms
Brief Title: Evaluating Pediatric Ivermectin in Children Under 15 kg (EPIC-15)
Acronym: EPIC-15
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other); Fundação de Dermatologia Tropical e Venereologia Alfredo da Matta (FUAM) (Unknown); University of Basel (Other); ClinSearch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAR22001
Record Dates: First submitted 2023-11-10; First posted 2024-05-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Scabies
Keywords: ivermectin; pediatric; CHILD-IVITAB
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (200 µg/kg) (Experimental)
  Interventions: Drug: CHILD-IVITAB
- Ivermectin (400 µg/kg) (Experimental)
  Interventions: Drug: CHILD-IVITAB

INTERVENTIONS:
Drug: CHILD-IVITAB — Ivermectin (200 µg/kg) oro-dispersible minitablets
  Arms: Ivermectin (200 µg/kg)
Drug: CHILD-IVITAB — Ivermectin (400 µg/kg) oro-dispersible minitablets
  Arms: Ivermectin (400 µg/kg)

SUMMARY:
The EPIC-15 trial will evaluate the safety, pharmacokinetics, acceptability, and efficacy of pediatric ivermectin (CHILD-IVITAB) in scabies infected children weighing 5 to less than 15 kg. This trial will support future efforts to expand the indication of ivermectin treatment to infants weighing 5 to less than 15 kg to treat numerous NTDs, allowing this young age group equitable access to the numerous benefits of pediatric ivermectin therapy

ELIGIBILITY:
Inclusion Criteria:

* Male or female child weighing 5 to <15 kilograms
* ≥3 months old
* Scabies infestation
* Available to attend all study visits
* Parents/guardians/carers able to provide written informed consent

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* A history of renal or hepatic impairment.
* Any other significant disease or disorder (e.g. moderate or severe malnutrition) which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who are participating or have participated in another research trial involving an investigational product in the past 12 weeks.
* Children with Crusted/Norwegian scabies or severe secondary bacterial infections (e.g. sepsis)
* Children who have taken ivermectin within the last month
* Children with known allergies to ivermectin or excipients
* Loa loa infection risk, assessed based on travel history to endemic areas
* Use of prescription (especially CYP3A4 inhibitors or inducers) or non-prescription drugs (except paracetamol at doses of up to 90 milligrams/kg/day), including vitamins (especially vitamin C), herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise participants safety; the investigator will take advice from the manufacturer representative as necessary.
* The investigator, health care provider or study staff feel that the participant is not suitable for study participation due to chronic illness, suspected underlying illness, or concerns that the participant will not adhere to follow-up schedule.
* Being born prematurely.
* Previously enrolled into this study

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Population pharmacokinetic properties of ivermectin concentrations at escalating doses in children <15 kg | Days 0, 3, 7, 10, 14

SECONDARY OUTCOMES:
Safety of oral ivermectin measures by pruritus outcomes assessed by a composite score recorded on the diary cards. | Assessments will be performed at planned visits on days 0, 3, 7, 10, 14, and daily via diary cards.
  Pruritus outcomes assessed by a composite score based on the behaviors displayed by the children as recorded on the diary cards.
Safety of oral ivermectin measures by percentage of children with abnormal biochemistry laboratory value | Assessments will be performed at planned visits on days 0, 3, 7, 10, 14
  Biochemistry laboratory value, including Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT), creatinine, and total bilirubin.
Safety of oral ivermectin measures by percentage of children with abnormal hematology laboratory value | Assessments will be performed at planned visits on days 0, 3, 7, 10, 14
  Hematology laboratory value including white blood cells, platelets, neutrophils, lymphocytes reported, hemoglobin, and hematocrit
Safety of oral ivermectin as measured by percentage of children with abnormal neurological test result. | Assessments will be performed at planned visits on days 0, 3, 7, 10, 14.
  Neurological test assesses by responses to a battery of stimuli with responses recorded as normal or abnormal.
Acceptability of pediatric oral ivermectin assessed by score of assessment tools called ClinSearch Acceptability Score Test (CAST) | Days 0, 7
  ClinSearch Acceptability Score Test (CAST) reports a barycenter and its 90% confidence ellipses on a 3D-map to assess positive
Efficacy of pediatric oral ivermectin to treat scabies in children <15 kg as measured by scabies lesion counts | Days 0, 7, 14

OTHER OUTCOMES:
Pharmacogenomics of ivermectin | Day 0
  Whole genome sequencing of study participants will be performed and related to safety, pharmacokinetics, and treatment efficacy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz von Seidlein, Dr, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Fundação de Dermatologia Tropical e Venereologia Alfredo da Matta (FUAM), Manaus, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: After publication
Access Criteria: Study data can be requested from the MORU Data Access Committee.